CLINICAL TRIAL: NCT05311345
Title: Integration of Cryobiopsies for ILD Diagnoses- Experience Based on 250 Biopsy Procedures.
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Sissel Kronborg-White, MD, principal investigator, Aarhus University Hospital
Organization: University of Aarhus (Other)
Other Study IDs: Cryobiopsy 250
Record Dates: First submitted 2020-04-17; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Interstitial Lung Disease
Keywords: Cryobiopsy
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective study on safety and Diagnostic yield in using cryobiopsies as a Diagnostic tool in diagnosing patients under investigation for Interstitial lung diseases. This includes a registration of procedural techniques, complications ( pneumthorax, hemorrhage, exacerbation and mortalt), days admitted at the hospital, diagnoses and diagnostic yield.

ELIGIBILITY:
Inclusion Criteria:

* >18years of age
* suspected of Interstitial lung Disease
* cryobiopsies performed.

Exclusion Criteria:

* FVC below 50% of predicted
* DLCO below 35%
* Body Mass Index (BMI) above 35
* pulmonary hypertension with a tricuspidal gradient above 40 mmHg
* other cardiac or other comorbidities that would increase the risk of complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under investigation for Interstitial lung diseases that were having cryobiopsies performed.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Pneumothorax | 2 weeks
  Pneumothorax, hemorrhage, acute exacerbation and death
Hemorrhage | 3 days
  Hemorrhage during the procedure
Acute exacerbation | 100 days
  Acute exacerbation after the procedure
Mortality | 100 days
  Mortality after the procedure

SECONDARY OUTCOMES:
Diagnostic yield | 1 month
  Diagnostic yield is discussed at multidisciplinary team meetings i.e, adequate biopsies (>50% alveolated biopsies), histologic pattern, kontribution to the diagnosis.

IPD SHARING:
Plan to Share IPD: Undecided
Participant data and study Protocol can be shared with other researcher upon reasonable request.